CLINICAL TRIAL: NCT02936336
Title: The Effect of Exercise Intervention on the Physical Fitness, Bone Mineral Density and Health-related Quality of Life in the Community's Older Adults
Brief Title: The Effect of Exercise Intervention on the Community's Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Robert Wen-Wei Hsu, Honorary Dean, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CMRPG690111-3;CMRPG6A0421-22
Record Dates: First submitted 2016-10-13; First posted 2016-10-18 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Metabolic Disease
MeSH Terms: conditions — Metabolic Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): without exercise intervention
- Exercise (Experimental): Subjects with circuit exercise, aerobic dance, or Tai Chi exercise intervention.
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — circuit exercise, aerobic dance and Tai Chi exercise
  Arms: Exercise

SUMMARY:
Osteoporosis is a serious global health problem, second only to cardiovascular disease. Osteoporosis is the most common metabolic bone disease in the elderly population, characterized by loss of bone mineral density (BMD) and continuous destruction of bone microstructure, especially in postmenopausal women. It gives rise to bone fragility and fracture risk. Moreover, as people grow older, falls frequently occur with high severity, and nearly 35% to 45% of persons aged 65 or older fall at least once a year. Osteoporotic fractures increase mortality, morbidity, chronic pain, and the cost of social care and it decreases the quality of life. Here, investigators plan to perform different exercise interventions such as circuit exercise, aerobic dance and Tai Chi on the community's older adults to evaluate whether exercise intervention could improve the bone mineral density, physical fitness, muscle strength or quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being >45 years-of-age,
* Healthy and physically independent.

Exclusion Criteria:

* The exclusion criteria were individuals on hormone replacement therapy and those with cognitive impairment, progressive debilitating conditions, bone fractures, or any medical contraindications to administering the fitness assessment.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2009-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline bone mineral density | Pre-intervention, 3-month, 6-month, 9-month-follow-up
  Bone mineral density measurement is measured by dual-energy x-ray absorptiometry (DXA). Measurements are made over the lumbar spine and over the upper part of the hip and the measurement is assessed at Pre-intervention, 3-month, 6-month, 9-month-follow-up.

SECONDARY OUTCOMES:
Change from baseline elbow muscle strength | Pre-intervention, 3-month, 6-month, 9-month-follow-up
  Extension and flexion of elbow were tested by the HUMAC NORM system (CSMi, Stoughton, MA) with the eccentric/concentric contraction mode at an angular velocity of 60 degrees/s.Isokinetic tests were performed five times for each participant, and each test was separated by a rest period of 3 min.The Muscle strength was present as a peak torque which was normalized to body weight (Unit:Nm/kg). The participants are assessed at Pre-intervention, 3-month, 6-month, 9-month-follow-up.
Change from baseline shoulder muscle strength | Pre-intervention, 3-month, 6-month, 9-month-follow-up
  Extension and flexion of shoulder were tested by the HUMAC NORM system (CSMi, Stoughton, MA) with the eccentric/concentric contraction mode at an angular velocity of 60 degrees/s.Isokinetic tests were performed five times for each participant, and each test was separated by a rest period of 3 min.The Muscle strength was present as a peak torque which was normalized to body weight (Unit:Nm/kg). The participants are assessed at Pre-intervention, 3-month, 6-month, 9-month-follow-up.
Change from baseline hip muscle strength | Pre-intervention, 3-month, 6-month, 9-month-follow-up
  Extension and flexion of hip were tested by the HUMAC NORM system (CSMi, Stoughton, MA) with the eccentric/concentric contraction mode at an angular velocity of 60 degrees/s.Isokinetic tests were performed five times for each participant, and each test was separated by a rest period of 3 min.The Muscle strength was present as a peak torque which was normalized to body weight (Unit:Nm/kg). The participants are assessed at Pre-intervention, 3-month, 6-month, 9-month-follow-up.
Change from baseline knee muscle strength | Pre-intervention, 3-month, 6-month, 9-month-follow-up
  Extension and flexion of knee were tested by the HUMAC NORM system (CSMi, Stoughton, MA) with the eccentric/concentric contraction mode at an angular velocity of 60 degrees/s.Isokinetic tests were performed five times for each participant, and each test was separated by a rest period of 3 min.The Muscle strength was present as a peak torque which was normalized to body weight (Unit:Nm/kg). The participants are assessed at Pre-intervention, 3-month, 6-month, 9-month-follow-up.
Change from baseline SF-36 questionnaire assessment | Pre-intervention, 3-month, 6-month, 9-month-follow-up
  SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower score the more disability. The higher the score the less disability. Eight sections including physical function, role limitation due to physical problems, bodily pain, general health, vitality, social functioning, role limitation due to emotional problems, and mental health. Additionally, the eight health domains can be used to provide a physical component summary and mental component summary score. The outcome measurement is assessed at Pre-intervention, 3-month, 6-month, 9-month-follow-up.
High-density lipoprotein from blood sample | Pre-intervention, 3-month, 6-month, 9-month-follow-up
  High-density lipoprotein are measured at Pre-intervention, 3-month, 6-month, 9-month-follow-up.
Triglyceride from blood sample | Pre-intervention, 3-month, 6-month, 9-month-follow-up
  Triglyceride are measured at Pre-intervention, 3-month, 6-month, 9-month-follow-up.
Fasting blood glucose from blood sample | Pre-intervention, 3-month, 6-month, 9-month-follow-up
  Fasting blood glucose are measured at Pre-intervention, 3-month, 6-month, 9-month-follow-up.
Blood pressure | Pre-intervention, 3-month, 6-month, 9-month-follow-up
  Diastolic and systolic blood pressure are measured at Pre-intervention, 3-month, 6-month, 9-month-follow-up.
Weight parameters of the subjects | Pre-intervention, 3-month, 6-month, 9-month-follow-up
  Weight (kg) are measured at Pre-intervention, 3-month, 6-month, 9-month-follow-up.
Height parameters of the subjects | Pre-intervention, 3-month, 6-month, 9-month-follow-up
  Height (cm) are measured at Pre-intervention, 3-month, 6-month, 9-month-follow-up.
Waistline parameters of the subjects | Pre-intervention, 3-month, 6-month, 9-month-follow-up
  Waistline (cm) are measured at Pre-intervention, 3-month, 6-month, 9-month-follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wen-Wei HSU, MD, Principal Investigator — Sports Medicine Center, Chang Gung Memorial Hospital, Chiayi
Locations (1):
- Sports Medicine Center, Chang Gung Memorial Hospital, Pizi, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hsu WH, Hsu WB, Fan CH, Hsu RW. Predicting osteoporosis with body compositions in postmenopausal women: a non-invasive method. J Orthop Surg Res. 2021 Mar 24;16(1):215. doi: 10.1186/s13018-021-02351-3. PMID 33761975